CLINICAL TRIAL: NCT06042270
Title: Thermoregulatory Responses of Betaine Supplementation in Firefighters During Live Burn
Brief Title: Firefighter Thermoregulatory Responses in Active Fire with Betaine Supplementation
Acronym: FFBET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael J. Ormsbee (Other)
Responsible Party: Sponsor-Investigator, Michael J. Ormsbee, Director, Florida State University
Organization: Florida State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00004218
Record Dates: First submitted 2023-08-25; First posted 2023-09-18 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-04

CONDITIONS: Body Temperature Changes; Body Water Dehydration; Inflammation
MeSH Terms: conditions — Body Temperature Changes; Dehydration; Inflammation | interventions — Betaine; Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 10 participants will be given rice-flour as a placebo
  Interventions: Dietary Supplement: Placebo
- Betaine (Active Comparator): 10 participants will be given betaine
  Interventions: Dietary Supplement: Betaine

INTERVENTIONS:
Dietary Supplement: Betaine — 3 grams per day for ~4 weeks
  Other Names: Trimethylglycine; Betaine Anhydrous
  Arms: Betaine
Dietary Supplement: Placebo — 3 grams per day for ~4 weeks
  Other Names: Rice Flour
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare betaine supplementation to placebo in firefighters undergoing live burn training regarding thermoregulation and inflammation. The main questions it aims to answer are:

* Does betaine supplementation mitigate rises in core temperature during firefighter live burn training?
* Does betaine supplementation decrease inflammation from firefighter training?
* Does betaine supplementation increase total body water stores?

Participants will supplement with betaine for 1 month and complete:

* Total Body Water measures
* Body Composition measures
* Live Burn training with Core Temperature Measurements
* Provide Salivary samples

ELIGIBILITY:
Inclusion Criteria:

* Structural Firefighter

Exclusion Criteria:

* • Participants have a cardiometabolic disease for which they take prescribed medications

  * Participants consume supplements known to impact hydration status or performance that they are not willing to stop taking for the study
  * Participants are pregnant
  * Female participants that have irregular menstrual cycles
  * Participants are injured and would not be able to fulfill the live burn scenario
  * Participants have sickle cell disease
  * Participants have experienced heat stroke within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Thermoregulation | 10 minutes before the live burn, during the ~15 minute live burn, 10, 20, and 30 minutes after the live burn.
  Core temperature (Degrees C), skin temperature (Degrees C)
Stress (enzyme linked immunoassays) | before, immediately after, 10 minutes, and 20 minutes after live burn
  Salivary expression of Testosterone, Cortisol, interleukin-8, and interleukin 6 will be measured.
Stress (respiration efficiency) | immediately before and immediately after the completion of the live burn
  Air tank pounds per square inch (PSI) will be recorded
Sweat Rate | immediately before and immediately after the completion of the live burn
  Changes in body weight in kg will be used to find loss of sweat in L
Sweat Content | immediately before and immediately after the completion of the live burn
  Tegaderm patches will be worn during the live burn to analyze sodium concentration in sweat.
Subjective measures | immediately before and immediately after the completion of the live burn
  Visual analog scales will be given to participants for subjective thermal sensation, rate of perceived exertion, and thirst

SECONDARY OUTCOMES:
Chronic Stress (enzyme linked immunoassays) | Before supplementation and after 4 weeks of supplementation
  Saliva will be analyzed for testosterone, cortisol, uric acid, and c-reactive protein
Chronic Stress (vitals) professional firefighters. | Before supplementation and after 4 weeks of supplementation
  Resting blood pressure in mmHg and heart rate in beats per minute will be measured.
Fluid Compartment Volumes (Bioelectrical Impedance Spectrocopy) professional firefighters. | Before supplementation and after 4 weeks of supplementation
  Intracellular fluid volume (L), extracellular fluid volume (L), plasma volume (L), total body water (L)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Science and Medicine, Tallahassee, Florida, United States